CLINICAL TRIAL: NCT01770054
Title: Evaluation of the Prevalence of Metabolic Syndrome in Atahualpa Residents Aged 40 Years or More.
Brief Title: Prevalence of Metabolic Syndrome in Atahualpa
Status: Completed | Type: Observational
Sponsor: Hospital Clínica Kennedy (Other)
Responsible Party: Principal Investigator, Oscar H. Del Brutto, MD, Rsearch Proffesor, Universidad de Especialidades Espiritu Santo, Hospital Clínica Kennedy
Other Study IDs: TAP 001-2013; 001-2013-01 (Other Grant/Funding Number: Universidad de Especialidades Espiritu Santo)
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; diabetes mellitus
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- obtention of a blood sample: all Atahualpa residents aged 40 years or more
  Interventions: Other: obtention of a blood sample

INTERVENTIONS:
Other: obtention of a blood sample — a blood sample will be obtained to measure glucose, HDL cholesterol, triglycerides, and for genetic testing

SUMMARY:
A recent epidemiologic survey demonstrated a high prevalence of type 2 diabetes mellitus in Atahualpa residents. Now, the investigators attempt to evaluate the prevalence of the metabolic syndrome in adults aged 40 years or more living in this rural village of coastal Ecuador.

DETAILED DESCRIPTION:
Several studies have shown that the occurrence of the metabolic syndrome is a risk factor for the development of cerebrovascular and ischemic heart disease. To evaluate the prevalence of the metabolic syndrome, we will invite all Atahualpa residents aged 40 years or more to participate in this study. For the purposes of this study we will obtain the waist circumference of all individuals, will measure their blood pressure using a standard protocol, and will take a blood sample to determine fasting glucose levels, HDL cholesterol levels, triglyceride levels, and plasma insulin levels.

ELIGIBILITY:
Inclusion Criteria:

* Atahualpa resident aged 40 years or more

Exclusion Criteria:

* non-consenting persons

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all Atahualpa residents aged 40 years or more
Sampling Method: Non-Probability Sample
Enrollment: 517 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of metabolic syndrome | 5 months
  determination of the metabolic syndrome in subjects aged 40 years or more

SECONDARY OUTCOMES:
Genetic testing | 5 months
  Blood will be taken to evaluate the ADN pattern of this population, to compare with other Amerindian populations with a proven high prevalence of diabetes mellitus and metabolic syndrome

OTHER OUTCOMES:
determination of the prevalence of hyperinsulinemia | 5 months
  plasma insulin levels will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Oscar H Del Brutto, MD, Principal Investigator — Universidad de Especialidades Espiritu Santo
Locations (1):
- Center of Health, Atahualpa, Santa Elena, Ecuador